CLINICAL TRIAL: NCT00283777
Title: Effect of Chromium Picolinate on Metabolic and Physiologic Parameters in Type 2 Diabetes
Brief Title: Chromium and Insulin Action
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, William Cefalu, MD, Executive Director, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 23041
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes
Keywords: insulin; glucose; body weight; chromium
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Body Weight | interventions — picolinic acid

INTERVENTIONS:
Drug: Chromium Picolinate

SUMMARY:
The effect of Chromium to improve glucose levels in diabetes is controversial. The hypothesis of the study was to evaluate the effect of supplementing the diet of individuals with Type 2 diabetes with chromium picolinate and assessing the effect on blood glucose levels and insulin sensitivity

DETAILED DESCRIPTION:
The primary clinical strategy to improve metabolic control in patients with Type 2 diabetes consists of lifestyle modification combined with pharmacologic intervention. However, alternative strategies, e.g. nutritional supplementation with over-the-counter agents, are extensively practiced by a large number of patients and are frequently undertaken without first informing the medical provider. Unfortunately, considerable controversy exists regarding use of dietary supplements in subjects with diabetes because efficacy data for many of the supplements consists of only uncontrolled studies and anecdotal reports. As such, there is a paucity of data in humans in regard to the effect of most commercially available supplements to improve metabolic abnormalities.

One supplement that has attracted considerable clinical interest is chromium (Cr). However, routine use of Cr in subjects with diabetes is not currently recommended. In part, the controversy surrounding Cr supplementation stems from the lack of definitive randomized trials, the lack of "gold standard" techniques to assess glucose metabolism in the studies reported, the use of differing doses and formulation , and the study of heterogeneous study populations (4). As such, conflicting data has been reported that has contributed greatly to the confusion among healthcare providers concerning Cr supplementation. In order to provide a comprehensive clinical evaluation of Cr, we conducted a randomized, double-blinded, placebo-controlled trial in subjects with Type 2 diabetes, and over a 10 month period of observation, used established techniques to assess changes in insulin sensitivity, body composition and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes on diet therapy or low dose oral agent -

Exclusion Criteria:

Significant cardiovascular, hepatic or renal disease

-

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1998-08; Primary Completion 2003-01 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Insulin Senstivity, glycated hemoglobin

SECONDARY OUTCOMES:
weight, body composition

CONTACTS AND LOCATIONS:
Overall Officials: William Cefalu, MD, Principal Investigator — University of Vermont and Pennington Biomedical Research Center
Locations (1):
- University of Vermont, Burlington, Vermont, United States